CLINICAL TRIAL: NCT01707069
Title: A Safety and Immunogenicity Phase I Study of CryJ2-DNA-Lysosomal Associated Membrane Protein (CryJ2 -DNA-LAMP) Plasmid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunomic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHI-2012
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Allergic Rhinoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: 4mg CryJ2-DNA-LAMP plasmid vaccine (Experimental): Healthy male and female subjects 18 to 63 years of age, who are skin test negative to Japanese Red Cedar pollen or Mountain Cedar pollen and have no reactive Cry J 2 antibodies.
  Group 1: will receive 4mg of Biological/Vaccine: CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection (considered to be the optimal DNA vaccine dose based on historical clinical data from other DNA vaccine studies). The dosing regimen for this group will be to receive three (3) additional booster doses (4 doses in total) of a 4 mg dose at 14 day intervals.
  Interventions: Biological: CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection
- Group 2: 2mg CryJ2-DNA-LAMP plasmid vaccine (Experimental): Healthy male and female subjects 18 to 63 years of age, who have lived in Japan, are Skin test positive to Japanese Red Cedar pollen or Mountain Cedar pollen and/or have reactive Cry J 2 antibodies, and have a history of allergic rhinitis symptoms during the Japanese Red Cedar or Mountain Cedar season will receive a total of four half (2 mg) dose dosing regimen.
  Group 2: will receive 2 mg Biological/Vaccine: CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection(considered ½ of the optimal plasmid vaccine dose based on historical clinical data from studies with other antigens). The dosing regimen for this group will be to receive three (3) additional 2 mg doses at 14 day intervals between doses (4 doses in total).
  Interventions: Biological: CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection
- Group 3: 4 mg CryJ2-DNA-LAMP plasmid vaccine (Experimental): Healthy male and female subjects 18 to 63 years of age, who have lived in Japan, are Skin test positive to Japanese Red Cedar pollen or Mountain Cedar pollen and/or have reactive Cry J 2 antibodies, and have a history of allergic rhinitis symptoms during the Japanese Red Cedar or Mountain Cedar season will receive a total of four full (4 mg) dose dosing regimen.
  Group 3: will receive 4 mg Biological/Vaccine: CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection (considered the optimal plasmid vaccine dose based on historical clinical data from studies with other antigens). The dosing regimen for this group will be to receive 3 additional 4 mg doses at 14 day intervals between doses (4 doses in total).
  Interventions: Biological: CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection

INTERVENTIONS:
Biological: CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection — Immunomic Therapeutics Inc. CryJ2-DNA-LAMP vaccine is a frozen product formulated in physiological saline and contains no preservative. The study product is packaged in a 1 ml volume in a 3 ml glass vial, with label complying with FDA requirements.
  Subjects will receive CryJ2-DNA-LAMP plasmid vaccine by intramuscular injection. The dosing regimen for this group will be to receive three (3) additional booster doses (4 doses in total) at 14 day intervals.

SUMMARY:
This is a research study of a vaccine for allergy to Japanese Red Cedar. The vaccine is called CryJ2-DNA-LAMP Plasmid vaccine. This research study will determine how the vaccine is tolerated and how research participants respond to the vaccine in various doses. CryJ2-DNA-LAMP Plasmid vaccine is investigational, which means it is not approved for use by the United States Food and Drug Administration (FDA) but is available in research studies like this one. This is the first time that CryJ2-DNA-LAMP Plasmid vaccine is being given to humans.

The purpose of this study is to evaluate the safety of an investigational vaccine intended to treat allergy to Japanese red cedar. The vaccine is composed of DNA, which is the material that cells use to provide instructions to make proteins. The DNA carries the information necessary to make a special protein which is a combination of a protein found in all cells, LAMP (lysosomal associated membrane protein), and the protein from Japanese red cedar that causes the allergy known as Cry J2. This vaccine is intended to help re-educate the immune system with respect to how it will respond to naturally occurring red cedar allergen and eliminate the allergic symptoms. Another purpose of this study will be to document the immune response to the vaccine

Subjects that are eligible to participate in this study will be assigned by whether they are sensitive or non sensitive to CryJ2 or Mountain Cedar and chance (like flipping a coin) to one of 3 study vaccine groups:

Group 1: will receive four (4) 4-milligram doses of the study vaccine. Group 2: will receive four (4) 2-milligram doses of the study vaccine. Group 3: will receive four (4) 4-milligram doses of the study vaccine.

The study vaccine is administered as an intramuscular injection. Enrolled subjects will receive the study vaccine every 14 days (at day 0, 14, 28 and 42). Subjects will know their study vaccine assignment. Participants who are not allergic to Japanese red cedar will be assigned to Group 1. Participants who do have an allergy to Japanese red cedar or Mountain Cedar will have an equal chance of being assigned to Group 2 or 3.

There will be between 18 to 30 men and women participating in the study at one location. Your participation in this study will last approximately 72 days.

DETAILED DESCRIPTION:
The study is a Phase I, prospective, three cohort, open label study conducted on one cohort of non-atopic subjects and two cohorts of patients with a history of allergic rhinitis symptoms to Japanese red cedar Cry j 2 pollen allergen. The study will be conducted at 1 study center. Subjects are enrolled in the trial for a period of 72 days. The objectives of the statistical analyses are to establish the safety and to explore the immunogenicity of the LAMP-vax vaccine. All statistical analyses conducted on the data from this trial will be exploratory in nature.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 and 63 years, are either:

   1. Japanese Red Cedar pollen or Mountain Cedar negative in skin tests and lack the presence of anti-Cry j 2 antibodies (To be assigned to Group 1)
   2. Japanese Red Cedar pollen or Mountain Cedar positive in skin tests and/or presence of anti-CryJ2 antibodies (to be assigned to Group 2 or 3).

      * For the purposes of this study, retrospective skin testing data (as long as it has been performed within 60 days of screening) will be accepted, using the same positive inclusion criteria
2. Execute a written informed consent (in English and where appropriate in Japanese) to participate in the study.
3. A minimum 1-year history of seasonal rhinoconjunctivitis (Nasal symptoms: sneezing, itching, rhinorrhea, congestion; Ocular symptoms: itching, redness, watering; Other: itching ears/throat) on exposure to Japanese Red Cedar pollen and/or Mountain Cedar pollen. Subjects have a clinical history that includes symptoms of allergic rhinitis during the Japanese Red Cedar or Mountain Cedar season and when exposed to Japanese Red Cedar and/or Mountain Cedar pollen.
4. Documented allergy to Japanese Red Cedar pollen as demonstrated by a positive epicutaneous skin test for Japanese Red Cedar pollen or Mountain Cedar antigen (wheal > 3mm greater than the negative control). Although, the subjects may have positive skin tests to other allergens, these will not be used to qualify or to participate in the study.
5. Female subjects of childbearing potential, defined as not surgically sterile or at least 2 years postmenopausal, must agree to use one of the following forms of contraception for the duration of the study: hormonal (oral, implant, or injection) begun >30 days prior to screening, barrier (condom, diaphragm with spermicide), intrauterine device (IUD), or vasectomized partner (6 months minimum).
6. No clinically significant abnormal findings on the physical examination, with the exception of HEENT findings consistent with allergic rhinitis, medical history, or clinical laboratory results during screening which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
7. Subject must be willing and able to comply with study requirements.

Exclusion Criteria:

1. Previous Japanese red cedar allergen immunotherapy (SCIT, oral immunotherapy, SLIT, or recombinant peptide)
2. History of anaphylaxis requiring medical intervention.
3. Intolerance of or severe allergic reaction to previous immunotherapy (SCIT, oral immunotherapy, SLIT, or recombinant peptide
4. History of asthma requiring daily medication with the exception of exercise induced asthma. (history of intermittent and/or mild asthma permitted)
5. Subjects receiving anti-IgE monoclonal antibodies.
6. Congenital immune deficiency or acquired immune suppression. Causes of acquired immune suppression may include, but are not limited to, systemic illnesses such as malignancy and infection, the use of medications such as corticosteroids and chemotherapeutic agents, and radiation therapy.
7. History of organ transplant, hematologic malignancy, autoimmune disease, myocardial infarction, or congestive heart failure.
8. History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic diseases, in the opinion of the Principal Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
9. Inability or unwillingness to stop using drugs that may inhibit the ability to treat a severe allergic adverse event. This includes, but is not limited to; beta blockers such as atenolol (Tenormin), metoprolol (Lopressor, Toprol-XL) and propranolol (Inderal, Inderal LA) for 48 hours prior to Visit 1 and for the duration of the study. All subjects must be off of antihistamine therapy 7 days before skin testing.
10. Female subjects who are trying to conceive, are pregnant, or are lactating.
11. Positive serum pregnancy test at screening or a positive human chorionic gonadotropin (HCG) urine test on Visit 1 for women of childbearing potential.
12. Positive blood screen for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbSAg), or Hepatitis C.
13. FEV1 of <70% as measure by spirometry.
14. Chronic history of recurrent sinusitis, urticaria or angioedema within the last 12 months.
15. History of alcohol or drug abuse within the year prior to the Screening Visit 1, or current evidence of substance dependence or abuse.
16. Laboratory Values (hematology, biochemistry, urine tests, PFT) that are outside the normal ranges, unless the abnormality is not considered clinically significant by the investigator.
17. Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to the Screening Visit.
18. Subjects with anti-LAMP antibodies above the Cutpoint Assay baseline will be excluded.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 72 days
  The primary objective of this Phase I Study is to evaluate the safety and immunological responses of therapeutic doses and the dosing regimen of CryJ2-DNA-LAMP plasmid vaccine.
  Adverse events will be monitored on each subject from the time of enrollment to exit from the study. Vital signs will be recorded on each subject at baseline and days 14, 28, 42 and 72. Clinical laboratory parameters will be obtained from blood samples taken at the baseline and final time points. Physical exams will be conducted on the subjects at the baseline and final time points.

SECONDARY OUTCOMES:
Immunogenicity and functional vairables | 72 days
  Immunogenicity parameters will be measured at baseline and days 14, 28, 42 and 72 or ET of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Fitz-Patrick, MD, Principal Investigator — East East Medical Research Institute
Locations (1):
- East West Medical Research Institute, Honolulu, Hawaii, United States